CLINICAL TRIAL: NCT05369182
Title: Prospective Registry of Coronary Flow-Derived Indexes in Patients With Coronary Artery Disease
Brief Title: Multicenter Registry of Coronary Flow-Derived Indexes for Coronary Microvascular Disease (Multicenter FLOW-CMD Registry)
Status: Active, not recruiting | Type: Observational
Sponsor: Samsung Medical Center (Other)
Collaborators: Chonnam National University Hospital (Other); Chosun University Hospital (Other); Seoul National University Bundang Hospital (Other); Seoul St. Mary's Hospital (Other)
Responsible Party: Principal Investigator, Joo Myung Lee, Professor, Samsung Medical Center
Other Study IDs: MulticenterFLOW
Record Dates: First submitted 2022-04-23; First posted 2022-05-11 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Coronary Microvascular Disease; Coronary Artery Disease; Ischemic Heart Disease
Keywords: Coronary Microvascular Disease; Coronary Artery Disease; Ischemic Heart Disease; Coronary Flow Reserve; Index of Microcirculatory Resistance; Fractional Flow Reserve; Intravascular Ultrasound; Optical Coherence Tomography
MeSH Terms: conditions — Microvascular Angina; Coronary Artery Disease; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Total Population: Patients with CMD (CFR<2.0 and IMR≥25): Among the enrolled patients, those who are diagnosed with CMD (CFR<2.0, IMR≥25) in physiologic assessment.
  Interventions: Diagnostic Test: Invasive physiologic assessment
- Total Population: Patients with preserved microvascular function (CFR≥2.0 OR IMR<25): Among the enrolled patients, those who are with preserved microvascular function (CFR≥2.0 OR IMR<25) in physiologic assessment.
  Interventions: Diagnostic Test: Invasive physiologic assessment
- Revascularized Population: Patients treated by intravascular imaging-guided PCI optimization: Among patients who received PCI, patients whose PCI was optimized through intravascular imaging device (IVUS or OCT).
  Interventions: Diagnostic Test: Invasive physiologic assessment; Diagnostic Test: Intravascular imaging
- Revascularized Population: Patients treated by angiography-only guided PCI: Among patients who received PCI, patients whose PCI was optimized through angiography-only.
  Interventions: Diagnostic Test: Invasive physiologic assessment

INTERVENTIONS:
Diagnostic Test: Invasive physiologic assessment — All coronary physiologic parameters are measured following diagnostic angiography. Resting pd/pa, FFR, CFR and IMR will be calculated using coronary physiologic parameters.
  In patients treated by PCI, post-PCI physiologic assessment including CFR, IMR, and FFR will be performed.
Diagnostic Test: Intravascular imaging — By the operator's discretion, stent-optimization will be performed under intravascular imaging devices (IVUS [Boston Scientific, Natick, Massachusetts, USA] or OCT [Abbott Vascular], St. Paul, MN, USA]).
  Groups: Revascularized Population: Patients treated by intravascular imaging-guided PCI optimization

SUMMARY:
Multicenter FLOW-CMD registry is a prospective, multi-center, registry study.

The aim of the study is to evaluate prognostic implications of coronary microvascular disease (CMD) in patients with ischemic heart disease (IHD) undergoing revascularization decision using FFR or other non-hyperemic pressure ratios.

DETAILED DESCRIPTION:
The diagnostic and therapeutic strategies in patients with coronary artery disease (CAD) have focused on identifying and alleviating both extent and severity of myocardial ischemia, as it is the most important prognostic fator. Thus, fractional flow reserve (FFR) has been a standard method for identifying ischemia-related epicardial coronary stenosis, accruing an abundance of clinical evidence on the benefit of FFR-guided treatment decisions. However, a high FFR value (>0.80) does not necessarily imply freedom from future events. Indeed, clinical events still occur in patients who are deferred based on high FFR. The microvasculature is one of the main components of coronary circulatory system, and the presence of microvascular disease may contribute to clinical events in patients without epicardial coronary stenosis. In the cardiac catheterization laboratory, microvascular disease can be assessed using a pressure/temperature-sensor coronary wire or a Doppler wire. Previous studies have demonstrated the incremental prognostic implications of coronary flow reserve (CFR) and index of microcirculatory resistance (IMR) in patients with high FFR, and the recent European guidelines supported the importance of invasive physiologic assessment using CFR and IMR in patients with stable coronary artery disease. Furthermore, recent Expert Consensus Documents and the European Society of Cardiology guideline of Chronic Coronary Syndrome have underlined the importance of evaluating coronary microvascular disease (CMD) in patients with ischemic heart disease (IHD) and proposed an universal definition of CMD based on: 1) functionally non-obstructive CAD defined by a fractional flow reserve (FFR)>0.80 and 2) impaired coronary microvascular function determined by abnormal CFR and/or microvascular resistance.

Another important issue in contemporary practice is how to improve patient prognosis after percutaneous coronary intervention (PCI). Although PCI can induce secondary CMD originated from multiple mechanism associated with the procedure (e.g. distal embolization or endothelial dysfunction), and although secondary CMD also affects coronary circulatory function, there has been no previous evidence evaluating the incidence and prognosis of secondary CMD after successful PCI for epicardial coronary stenosis. Furthermore, both previous and recent trials demonstrated that intravascular imaging-guided PCI optimization has significantly better clinical outcomes than angiography-only guided PCI. However, these trials could not explain the exact mechanism underlying the potential benefit of intravascular imaging-guided PCI optimization for better clinical outcome, aside from a larger final stent area following intravascular imaging-guided PCI. Although the fundamental purpose of PCI is to resolve inducible myocardial ischemia originated from epicardial coronary stenosis, several studies have demonstrated that a substantial proportion of patients who underwent angiographically successful PCI had suboptimal post-PCI FFR or non-hyperemic pressure ratios, which are independently associated with worse clinical outcomes. Previous studies demonstrated that intravascular imaging devices could identify correctable cause of suboptimal post-PCI FFR. In this regard, it can be expected that intravascular imaging-guided PCI optimization would result in better post-PCI physiologic results such as higher post-PCI FFR and CFR, compared with angiography-only guided PCI.

However, these issues have not been fully clarified. Regarding the prognostic impact of CMD, only limited data has been available on the prognostic implications of CMD defined by the universal definition among patients with IHD, especially in patients with insignificant epicardial coronary disease defined by FFR>0.80. In addition, only one prospective study evaluated optical coherence tomography (OCT)-guided PCI for post-PCI FFR in patients with non-ST segment elevation myocardial infarction. None of prospective study evaluated potential physiologic benefit of intravascular imaging-guided PCI optimization using intravascular ultrasound (IVUS) or OCT in unselected patient population.

Therefore, the primary objectives of the current multicenter prospective registry are to evaluate prognostic implications of CMD in patients with suspected IHD undergoing revascularization decision using FFR or other non-hyperemic pressure ratios and to evaluate the efficacy of intravascular imaging-guided optimization to enhance post-revascularization coronary circulatory function, compared with angiography-only guided revascularization in revascularized population.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be ≥18 years
2. Patients suspected with IHD
3. Patients undergoing physiologic assessment (CFR, IMR, and FFR) for evaluation of severity of CAD
4. Subject is able to verbally confirm understandings of risks, benefits and treatment alternatives of receiving invasive physiologic or imaging evaluation and he/she or his/her legally authorized representative provides written informed consent to any study related procedure.

Exclusion Criteria:

1. Cardiogenic shock (systolic blood pressure <90mmHg or requiring inotropics to maintain blood pressure >90mmHg) or cardiac arrest
2. Non-cardiac co-morbid conditions are present with life expectancy <2 year (per site investigator's medical judgment).
3. Inability to undergo physiologic assessment (CFR, IMR, and FFR)
4. Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected IHD undergoing invasive coronary angiography and clinically indicated physiological assessment will be eligible. A total of 1,003 patients will be enrolled at 7 centers in South Korea.
Sampling Method: Non-Probability Sample
Enrollment: 1003 (Actual)
Dates: Start 2022-04-22 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient-oriented composite outcomes (POCO) | 1 year after last patient enrollment
  a composite of all-cause death, MI, any repeat revascularization, or admission for heart failure

SECONDARY OUTCOMES:
All-cause death | 1 year after last patient enrollment
  All-cause death
Cardiac death | 1 year after last patient enrollment
  Cardiac death
Target-vessel MI | 1 year after last patient enrollment
  Target-vessel MI
Non-target vessel MI | 1 year after last patient enrollment
  Non-target vessel MI
Any MI | 1 year after last patient enrollment
  Any MI
Target vessel revascularization (clinically-driven or all) | 1 year after last patient enrollment
  Target vessel revascularization (clinically-driven or all)
Non-target vessel revascularization (clinically-driven or all) | 1 year after last patient enrollment
  Non-target vessel revascularization (clinically-driven or all)
Any repeat revascularization (clinically-driven or all) | 1 year after last patient enrollment
  Any repeat revascularization (clinically-driven or all)
Admission for congestive heart failure | 1 year after last patient enrollment
  Admission for congestive heart failure
Stroke (ischemic and hemorrhagic) | 1 year after last patient enrollment
  Stroke (ischemic and hemorrhagic)
Seattle Angina Questionnaire | Baseline, 1 year, and 2 year after patient enrollment
  Physical limitation, Angina stability, Angina frequency, Treatment satisfaction, Quality of life
Proportion of functionally optimized post-PCI results | Post-procedure
  Proportion of functionally optimized post-PCI results (Post-PCI FFR>0.80 and CFR>2.0) according to the use of intravascular imaging
Incidence of secondary CMD after PCI | Post-procedure
  Incidence of secondary CMD (CFR<2.0 and IMR≥25) after PCI among revascularized population

CONTACTS AND LOCATIONS:
Overall Officials: Joo Myung Lee, MD, MPH, PhD, Principal Investigator — Samsung Medical Center
Locations (7):
- South Korea (7):
  - Chonnam National University Hospital, Gwangju
  - Chosun University Hospital, Gwangju
  - Gyeongsang National University Hospital, Jinju
  - Seoul National University Bundang Hospital, Seongnam
  - Samsung Medical Center, Seoul
  - Seoul National University Boramae Medical Center, Seoul
  - Seoul St. Mary's Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Yes
After publication of first manuscript and trial results, the de-identified data will be shared by permission of principle investigator, when asked
Supporting Information: Study Protocol, CSR
Time Frame: After publication of first manuscript and trial results
Access Criteria: The de-identified data will be shared by permission of principle investigator, when asked